CLINICAL TRIAL: NCT03459703
Title: Effect of Time-Restricted Feeding on Fat Loss and Cardiometabolic Risk Factors in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Courtney M Peterson, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001207
Record Dates: First submitted 2018-02-14; First posted 2018-03-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: Statistical analyses will be performed blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time-Restricted Feeding (Experimental)
  Interventions: Behavioral: Early Time-Restricted Feeding; Behavioral: Structured Weight Loss Program
- Control Schedule (Active Comparator)
  Interventions: Behavioral: Control Schedule; Behavioral: Structured Weight Loss Program

INTERVENTIONS:
Behavioral: Early Time-Restricted Feeding — Eat all meals between 7 am - 3 pm for an average of ≥6 days per week.
  Other Names: Early TRF; eTRF
  Arms: Early Time-Restricted Feeding
Behavioral: Control Schedule — Eat all meals over a 12-hour or longer period for an average of ≥6 days per week.
  Arms: Control Schedule
Behavioral: Structured Weight Loss Program — A structured weight loss program with physical activity recommendations and dietary counseling.

SUMMARY:
Time-restricted feeding (TRF) is a novel type of intermittent fasting that involves eating within a daily period of 10 hours or less, followed by fasting for at least 14 hours daily. Several studies in rodents report that TRF reduces body weight, improves blood sugar control, and reduces the risk of cardiovascular disease-even when food intake is matched to the control group or no weight loss occurs. Preliminary evidence suggests that TRF may also increase weight loss, fat loss, and reduce the risk of diabetes and cardiovascular disease in humans. This study will test whether TRF enhances fat loss and increases weight loss in adults with obesity, relative to conventional dieting alone. In addition, this study will determine whether TRF reduces risk factors for type 2 diabetes and cardiovascular disease and will measure the feasibility and acceptability of TRF.

In conjunction with the parent study described above, four ancillary studies will be conducted:

1. Effect of weight loss on nitrogen metabolism and bacteria in the mouth. The primary endpoints for this ancillary study are plasma and salivary nitrate and nitrite, and the secondary endpoints are salivary nitrate reductase activity and salivary bacterial abundance.
2. Effect of weight loss on several biomarkers related to kidney stones. The primary endpoint for this ancillary study is urinary oxalate, and the secondary endpoints are urinary citrate, chloride, sodium, potassium, calcium, phosphorus, uric acid, and creatinine.
3. Effect of meal timing on blood pressure regulation and kidney function. The primary endpoints of this ancillary study include urinary aldosterone excretion, sodium, potassium, and endothelin, whereas the secondary endpoints include nitric oxide and albumin. Additional exploratory endpoints include renal injury markers (KIM-1, nephrin, and urine albumin-to-creatinine ratio), measures of reactive oxidative stress (e.g., hydrogen peroxide and TBARs), and urinary exosomes. Urine will be analyzed in 12-hour bins to determine how meal timing affects differentially affects these endpoints during the daytime and nighttime. The effects of weight loss on these endpoints may also be considered.
4. Validation of a meal timing questionnaire to assess the distribution of food intake throughout the day.

ELIGIBILITY:
Inclusion Criteria:

* Are a new patient at the UAB Weight Loss Medicine Clinic
* Aged 25-75 years old
* BMI between 30-60 kg/m2 (inclusive)
* Weigh less than 450 lbs
* Wake up regularly between 4-9 am on most days.

Exclusion Criteria:

* Diagnosed with diabetes, have an HbA1c of ≥6.5%, or are on diabetes medication
* On weight loss medication
* Addition of or withdrawal from a chronic medication within the past 10 weeks
* Clinically significant laboratory abnormality (e.g., abnormal hemoglobin levels)
* Significant gastrointestinal disease, major gastrointestinal surgery, or gallstones
* Significant cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that might compromise the participant's safety or data validity
* Evidence of cancer (other than non-melanoma skin cancer) within the last 5 years
* Unstable psychiatric, sleep, or circadian conditions (common conditions such as sleep apnea and depression are acceptable as long as they are stabilized and not rapidly worsening)
* Lost or gained more than 5 lbs of weight in the past month
* Currently perform overnight shift work more than once per week on average
* Regularly eat within a less than 10-hour period each day
* Regularly eat dinner before 6 pm
* Traveled more than two time zones away in the two months prior to enrolling in the trial
* Will travel more than one time zone away during the study
* Pregnant or breastfeeding

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Fat loss and lean mass retention | 14 weeks
  Percent of weight lost as fat, as measured by dual-energy X-ray absorptiometry (DXA). Lean mass retention will be quantified as 100% minus percent of weight lost as fat (i.e., is measured in the same units).
Weight loss | 14 weeks
  Change in body weight (kg), as measured by scale weight
Absolute changes in body composition | 14 weeks
  Changes in total fat mass, lean mass, bone mass, and regional values (kg), as measured by DXA. (This will be secondary to the assessment of fat loss and lean mass retention as specified above.)

SECONDARY OUTCOMES:
Fasting glucose | 14 weeks
  Fasting glucose (mg/dl)
Fasting insulin | 14 weeks
  Fasting insulin (IU/L)
HbA1c | 14 weeks
  HbA1c (%)
Lipids | 14 weeks
  Total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl)
Blood pressure | 14 weeks
  Systolic and diastolic blood pressure (mm Hg)
Heart rate | 14 weeks
  Heart rate in beats per minute
Waist circumference | 14 weeks
  Waist circumference (cm)

OTHER OUTCOMES:
Appetite | 14 weeks
  Hunger and fullness as measured by Likert (1-5 scale) and visual analog scales (a 0-100 scale, with 0 meaning "Not at all" and 100 meaning "Extremely")
Food intake | 14 weeks
  Energy intake and food intake in kcal/day, as measured using Remote Food Photography Method (RFPM)
Macronutrient intake | 14 weeks
  % of calories as fat, carbohydrate, and protein, as measured using RFPM
Meal frequency | 14 weeks
  Number of meals and snacks per day, as measured using RFPM
Meal times | 14 weeks
  Clock times of meals and snacks, as measured using RFPM
Times of eating | 14 weeks
  Start and stop times and mid-points of daily eating in clock time, as assessed by the daily adherence survey
Duration of daily eating | 14 weeks
  Average duration of the daily eating period (hours), as measured by the daily adherence survey
Distribution of food intake across the daytime | 14 weeks
  Distribution of calories eaten across the day in % per time period, as measured by a novel questionnaire that is being validated
Breakfast and nighttime eating habits | 14 weeks
  Presence and degree of breakfast and nighttime eating, as measured by a novel questionnaire that is being validated
Adherence | 14 weeks
  Self-reported adherence rate in days per week
Reasons for non-adherence | 14 weeks
  Reasons for non-adherence, as measured by the daily adherence survey
Retention | 14 weeks
  Attrition rate (%)
Depression | 14 weeks
  Depression as measured by the Patient Health Questionnaire-9. (Each question is scored on a 0-3 scale, where 0 means "Not at all" and 3 means "Nearly every day." Answers to each question are tallied to create a single composite score of depression from 0-27, with higher values meaning more depressive symptoms.)
Mood states | 14 weeks
  Mood states as measured by the Profile of Mood States (a 5-point scale with 1 meaning "Not at all" and 5 meaning "Extremely"). This study is particularly interested in the scores for anxiety and related moods.
Chronotype | 14 weeks
  Chronotype/mid-point of sleep (in clock time), as measured by the Munich Chronotype Questionnaire
Stimulant usage | 14 weeks
  Stimulant usage, as measured by the Munich Chronotype Questionnaire (in "servings" per time)
Sleep duration | 14 weeks
  Sleep duration, as measured by the Pittsburgh Sleep Quality Index
Sleep quality | 14 weeks
  Sleep quality, as assessed by the Pittsburgh Sleep Quality Index (PQSI) (This study will use the Global PQSI score, which ranges from 0-21, where higher values correspond to worse sleep quality.)
Eating Behaviors | 14 weeks
  Restrained, emotional, and external eating, as measured by the Dutch Eating Behavior Questionnaire. (Individual questions are scored on a 5-point scale ranging from "Never" to "Very often," and composite scores for restrained, emotional, and external eating are tabulated, with higher numbers reflecting more of each trait.)
Loneliness | 14 weeks
  Loneliness, as measured by the UCLA Loneliness Scale (a 3-point scale with 1 meaning "hardly ever" and 3 meaning "often")
Intervention satisfaction | 14 weeks
  Intervention satisfaction and barriers and facilitators of adherence, as measured by qualitative exit interview
Social life and daily habits | 14 weeks
  Social life and daily habits, as measured by the frequency of occurrence of social activities (5- and 8-point rating scales)
Physical activity | 14 weeks
  Physical activity status, as measured by the Baecke Physical Activity questionnaire
Plasma and salivary nitrate and nitrite | 14 weeks
  Plasma and salivary nitrate and nitrite (nM)
Salivary nitrate reductase activity | 14 weeks
  Salivary nitrate reductase activity (nmol / min / colony forming unit) in tongue swab samples
Salivary bacterial abundance | 14 weeks
  Salivary bacterial abundance (colony forming units) in tongue swab samples
24-hour urinary oxalate, citrate, sodium, calcium, chloride, potassium, and creatinine | 14 weeks
  24-hour urinary oxalate, citrate, sodium, calcium, chloride, potassium, and creatinine, as measured in mg/day
24-hour urinary phosphorus and uric acid | 14 weeks
  24-hour urinary phosphorus and uric acid, as measured in g/day
24-hour urinary aldosterone excretion | 14 weeks
  24-hour urinary aldosterone excretion (µg/12 hr)
12-hour urinary sodium and potassium | 14 weeks
  12-hour urinary sodium and potassium (mmol/12 hr)
12-hour urinary endothelin | 14 weeks
  12-hour urinary endothelin (ng/12 hr)
12-hour urinary nitric oxide | 14 weeks
  12-hour urinary nitric oxide (mmol/12 hr)
12-hour urinary albumin | 14 weeks
  12-hour urinary albumin (mg/12 hr)
12-hour urinary KIM-1 | 14 weeks
  12-hour urinary KIM-1 (pg/g creatinine or pg/12 hr)
12-hour urinary nephrin | 14 weeks
  12-hour urinary nephrin (ng/g creatinine or ng/12 hr)
12-hour albumin-to-creatinine ratio | 14 weeks
  12-hour albumin-to-creatinine ratio
12-hour urinary reactive oxidative stress | 14 weeks
  12-hour urinary hydrogen peroxide and TBARs (µmol/g creatinine or µmol/12 hr)
Urinary exosomes | 14 weeks
  Urinary exosomes (particles/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Peterson, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Weight Loss Medicine Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Jamshed H, Steger FL, Bryan DR, Richman JS, Warriner AH, Hanick CJ, Martin CK, Salvy SJ, Peterson CM. Effectiveness of Early Time-Restricted Eating for Weight Loss, Fat Loss, and Cardiometabolic Health in Adults With Obesity: A Randomized Clinical Trial. JAMA Intern Med. 2022 Sep 1;182(9):953-962. doi: 10.1001/jamainternmed.2022.3050. PMID 35939311
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717